CLINICAL TRIAL: NCT03510468
Title: Impact of Weekly Administration of Rifapentine and Isoniazid on Steady State Pharmacokinetics of Tenofovir Alafenamide in Healthy Volunteers
Brief Title: Impact of Weekly Administration of Rifapentine and Isoniazid on Steady State Pharmacokinetics of Tenofovir Alafenamide in Healthy Volunteers (YODA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 180087; 18-CC-0087
Record Dates: First submitted 2018-04-26; First posted 2018-04-27 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2022-12-21

CONDITIONS: Healthy Volunteers
Keywords: Antiretroviral Therapy; Human Immunodeficiency Virus; Latent Tuberculosis; Drug-Drug Interactions; Rifamycin
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Latent Tuberculosis | interventions — tenofovir alafenamide; rifapentine; Isoniazid; Pyridoxine; Vitamin B 6

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pharmacokinetic study in healthy volunteers (Experimental): Healthy volunteers received Tenofovir alafenamide (TAF) 25 mg once daily for 14 days followed by TAF 25 mg once daily and Rifapentine (RPT) dosed by weight in 150-mg tablet increments (maximum oral dose of 900 mg) 750 or 900 mg (depending on weight) and Isoniazid (INH+ pyridoxine), 15 mg/kg (up to 900 mg) once weekly from days 15-31.
  Interventions: Drug: Tenofovir alafenamide; Drug: Rifapentine; Drug: Isoniazid (INH); Dietary Supplement: Pyridoxine

INTERVENTIONS:
Drug: Tenofovir alafenamide — Each tablet contains 25 mg of tenofovir alafenamide.
  Other Names: Vemlidy
Drug: Rifapentine — Each tablet contains 150 mg of rifapentine. Participants who weigh 45 to < 50 kg will take 750 mg (5 tablets), and participants who weigh (Bullet) 50 kg will take 900 mg (6 tablets).
  Other Names: Priftin
Drug: Isoniazid (INH) — Each tablet is formulated as 100 or 300 mg of isoniazid.
Dietary Supplement: Pyridoxine — Each tablet contains 50 mg of pyridoxine
  Other Names: Vitamin B6

SUMMARY:
Background:

Human immunodeficiency virus (HIV) is treated with antiretroviral drugs. Many people with HIV also have the lung infection tuberculosis (TB). Most TB treatments are complicated. A simpler treatment of two TB drugs can be taken once a week. Researchers want to study how the HIV and TB drugs affect each other so people who take both can be treated safely.

Objective:

To study if rifapentine and isoniazid affect blood levels of the common antiretroviral TAF.

Eligibility:

Healthy adults ages 18-65 without HIV, TB, or hepatitis

Design:

Participants will fast before the screening visit. They will have a medical history, physical exam, and blood tests. Women may have a pregnancy test.

During the study, participants must:

Use effective birth control

Not take most medicine

Not drink alcohol

At the baseline visit, participants will repeat screening tests and get TAF tablets.

Participants will take TAF once a day for 31 days. They will keep track of doses and side effects.

Over 32 days, participants will have 4 long visits and 4 short.

At all visits, participants will:

Fast the night before

Get food

Take that day's TAF

Review their TAF supply

Have pregnancy and blood tests

Report side effects

At 3 visits, participants will also take the 2 TB drugs and vitamin B6.

At 3 long visits, participants will also have blood collected 8 times over 8 hours by plastic tube in an arm vein.

Around Day 46, participants will fast and have blood and pregnancy tests. Two weeks later, they will get a call to see how they are feeling.

DETAILED DESCRIPTION:
Rifapentine (RPT) is a long-acting rifamycin that can be used weekly with isoniazid (INH) as a first-line regimen in the treatment of latent tuberculosis infection (LTBI). Although this regimen offers several potential benefits, the use of weekly RPT plus INH is limited in adults infected with human immunodeficiency virus (HIV) on antiretroviral therapy (ART) due to lack of drug interaction data with antiretrovirals (ARVs). Tenofovir alafenamide (TAF) is a preferred backbone agent by the current Department of Health and Human Services ARV guidelines and is a part of multiple recommended first-line regimens for the treatment of HIV. However, the use of TAF with rifamycins, including RPT, is not recommended due to potential drug interactions. Thus, the purpose of this study is to determine the effects of concomitant RPT and INH administration on the steady state pharmacokinetics (PK) of plasma TAF, plasma tenofovir (TFV), and intracellular TFV diphosphate (dp).

This is an open-label, fixed sequence, intrasubject drug-drug interaction study designed to evaluate the steady state PK of TAF, TFV, and TFV-dp with coadministration of once-weekly RPT + INH administered at doses used to treat LTBI. The study will consist of two phases: (1) TAF once daily alone (days 1-14) and (2) TAF once daily + weight-based RPT + INH once weekly (days 15-31). Participants will undergo periodic serial ARV PK blood draws over 24 hours on days 14-15, 22-23, and 31-32.

TAF, TFV, and TFV-dp PK will be determined using non-compartmental methods. The following PK parameters will be compared between phases: area under the curve over the dosing interval, maximum plasma concentration, time to maximum plasma concentration, terminal half-life, apparent oral clearance, and minimum plasma concentration. Adverse events will be graded and recorded.

ELIGIBILITY:
* PARTICIPANT INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

1. Ages 18-65 years.
2. Weight greater than or equal to 45 kg and less than or equal to 120 kg OR body mass index greater than or equal to 18.0 and < 30.
3. Judged to be healthy based on medical history, physical examination, vital signs, and clinical laboratory tests: liver function tests (AST, alanine transaminase( ALT), Tbili) less than or equal to upper limit of normal [ULN], serum creatinine (SCr) less than or equal to ULN, platelets (PLT) > 150,000/microL, hemoglobin (Hgb) > 13 g/dL (males); greater than or equal to 12g/dL (females), C-reactive protein (CRP) less than or equal to ULN, creatine kinase (CK) less than or equal to 2x ULN, fasting total cholesterol < 240 mg/dL, or fasting triglycerides < 240 mg/dL, urine glucose < grade 2 (per Division of Acquired Immunodeficiency Syndrome (DAIDS) adverse event (AE) table), urine protein < grade 2 (per DAIDS AE table).
4. Negative QuantiFERON-TB Gold test at screening.
5. HIV-negative, as determined by standard serologic assays for HIV infection.
6. No laboratory evidence of active or chronic hepatitis A, B, or C infection.
7. Willing to abstain from alcohol consumption throughout the study period.
8. Agrees to genetic testing and storage of specimens for future research.
9. Able to provide informed consent.
10. Negative serum or urine pregnancy test for females of child-bearing potential.
11. Participants must agree not to become pregnant or impregnate a partner for the duration of the study. The use of hormonal contraceptives will not be permitted. Study participants must use one of the following methods of birth control when engaging in sexual activities that can result in pregnancy, beginning at screening until the final study visit.

    1. Male or female condom.
    2. Diaphragm or cervical cap with a spermicide.
    3. Intrauterine device without hormones.

PARTICIPANT EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

1. Known hypersensitivity to TAF, tenofovir disoproxil fumarate (TDF), INH, RPT, and other rifamycin analogues.
2. History or presence of any of the following:

   1. Latent or active TB infection.
   2. Gastrointestinal (GI) disease that is uncontrolled, requires daily treatment with medication, or would interfere with a participant s ability to absorb drugs (eg, diarrhea, pancreatitis, or peptic ulcer disease).
   3. Renal impairment (chronic renal insufficiency of any chronic kidney disease stage, or acute renal failure not induced by drug therapy defined as estimated glomerular filtration rate (eGFR) < 90 mL/min or SCr > ULN).
   4. Respiratory disease that is uncontrolled or requires daily treatment with medication (eg, asthma or chronic obstructive pulmonary disease).
   5. Cardiovascular disease (eg, hypertension [systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mm Hg], heart failure, or arrhythmia).
   6. Metabolic disorders (eg, diabetes mellitus).
   7. Hematologic or bleeding disorders (eg, anemia, hemophilia, serious/major bleeding events, menorrhagia [female participants]).
   8. Immunologic disorders.
   9. Hormonal or endocrine disorders.
   10. Psychiatric illness that would interfere with their ability to comply with study procedures or that requires daily treatment with medication.
   11. Seizure disorder, with the exception of childhood febrile seizures.
   12. Any current or history of malignancy, with the exception of cutaneous basal cell carcinoma,non-invasive squamous cell carcinoma, or any other malignancies not requiring systemic

       therapy.
   13. Current or history of osteopenia and osteoporosis.
3. Current participation in an ongoing investigational drug protocol or use of any investigational drug within 30 days (based on last dose received) prior to receipt of any study drugs.
4. Therapy with any prescription, over-the-counter (OTC), herbal, or holistic medications, including hormonal contraceptives by any route, within 5 half-lives of the agent prior to receipt of any study medications will not be permitted with the following exception: Intermittent or short-course therapy (<14 days) with prescription or OTC medications, herbals, or holistic medications within the screening period prior to starting study drugs may be permitted, and will be reviewed by investigators on a case-by-case basis for potential drug interactions. Receipt of influenza vaccination will be allowed prior to, during, and/or after the study.
5. Inability to obtain venous access for sample collection.
6. Inability to swallow whole capsules and/or tablets.
7. Pregnant or breastfeeding.
8. Drug use that may impair safety or adherence.
9. Use of nicotine-containing products, including cigarettes and chewing tobacco, nicotine patches, gum, electronic cigarettes, etc.
10. Organ or stem cell transplant recipient.
11. Uncorrected and persistent electrolyte abnormalities (eg, potassium, magnesium, and calcium).
12. Current alcohol use disorders (DSM-5 criteria).
13. Fasting total cholesterol > 240 mg/dL or fasting triglycerides > 240 mg/dL at screening.
14. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
.Individual participant data will not reported or shared. The study team are the only individuals who have access to individual participant data. All data will be analyzed and reported in aggregate.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-CC-0087.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 51 participants consented to the study, 17 were screen failure and 6 withdrew prior to start of study.
Period: Overall Study
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Started | 28
Completed | 18
Not Completed | 10
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 5
Not completed — Physician Decision | 1
Not completed — non-compliant with treatment | 2
Not completed — Missed visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 13
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Plasma Area Under the Curve (AUC) for Tenofovir Alafenamide (TAF) During the Dosing Interval of 0 to 24 Hours (AUC0-24hr)
Description: Plasma area under the curve (AUC) during the dosing interval of 0 to 24 hours (AUC0-24hr) on day 14, 22, and 31 of TAF was calculated using the linear-up/log-down trapezoidal rule using noncompartmental methods on Phoenix WinNonlin ®
Time Frame: 0-24 hours post dosing on days 14, 22, and 31
Population: All participants who completed at least one intensive pharmacokinetic visit were included in the pharmacokinetics analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 20
hr*ng/ml
  Day 14: number analyzed (Participants) | 19
  Day 14 | 295.5 (64)
  Day 22 | 472.1 (59)
  Day 31: number analyzed (Participants) | 16
  Day 31 | 248.1 (88)

2. Primary Outcome: Plasma Area Under the Curve (AUC) for Tenofovir (TFV) During the Dosing Interval of 0 to 24 Hours (AUC0-24hr)
Description: Plasma area under the curve (AUC) during the dosing interval of 0 to 24 hours (AUC0-24hr) on day 14, 22, and 31 of TFV was calculated using the linear-up/log-down trapezoidal rule using noncompartmental methods on Phoenix WinNonlin ®
Time Frame: 0-24 hours post dosing on days 14, 22, and 31
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 21
hr*ng/ml
  Day 14 | 262.2 (45)
  Day 22: number analyzed (Participants) | 20
  Day 22 | 265.3 (38)
  Day 31: number analyzed (Participants) | 15
  Day 31 | 230.8 (45)

3. Primary Outcome: Maximum Total Plasma Concentration (Cmax) for Tenofovir Alafenamide (TAF)
Description: Maximum total plasma concentration (Cmax) following a 25mg dose of TAF on day 14, 22, and 31. Cmax for TAF was obtained directly by visual inspection of the plasma concentration versus time profiles over 24 hours postdose.
Time Frame: Days 14, 22, and 31
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 23
ng/mL
  Day 14 | 208.9 (88)
  Day 22: number analyzed (Participants) | 22
  Day 22 | 335.2 (61)
  Day 31: number analyzed (Participants) | 16
  Day 31 | 179.1 (80)

4. Primary Outcome: Maximum Total Plasma Concentration (Cmax) for Tenofovir (TFV)
Description: Maximum total plasma concentration (Cmax) following a 25mg dose of tenofovir alafenamide (TAF) on day 14, 22, and 31. Cmax for TFV was obtained directly by visual inspection of the plasma concentration versus time profiles over 24 hours postdose.
Time Frame: Days 14, 22, and 31
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 22
ng/mL
  Day 14 | 16.5 (79)
  Day 22: number analyzed (Participants) | 20
  Day 22 | 16.5 (37)
  Day 31: number analyzed (Participants) | 15
  Day 31 | 13.8 (35)

5. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) for Tenofovir Alafenamide (TAF)
Description: Time to maximum total plasma concentration (Cmax) following a 25mg dose of TAF on day 14, 22, and 31. Tmax for TAF was obtained directly by visual inspection of the plasma concentration versus time profiles over 24 hours postdose.
Time Frame: Days 14, 22, and 31
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 23
Hours
  Day 14 | 0.5 [0.25 to 2]
  Day 22: number analyzed (Participants) | 22
  Day 22 | 0.57 [0.25 to 2]
  Day 31: number analyzed (Participants) | 16
  Day 31 | 0.5 [0.25 to 2]

6. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) for Tenofovir (TFV)
Description: Time to maximum total plasma concentration (Cmax) following a 25mg dose of TAF on day 14, 22, and 31. Tmax for TFV was obtained directly by visual inspection of the plasma concentration versus time profiles over 24 hours postdose.
Time Frame: Days 14, 22, and 31
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 22
Hours
  Day 14 | 4 [0.25 to 8]
  Day 22: number analyzed (Participants) | 20
  Day 22 | 4 [1 to 4.1]
  Day 31: number analyzed (Participants) | 15
  Day 31 | 4 [0 to 8]

7. Primary Outcome: Terminal Half-life (t½) of Tenofovir (TFV)
Description: Half-life calculated as natural log of 2 [ln(2)]/lambda Z of TFV on day 14, 22, and 31.
Time Frame: Days 14, 22, and 31
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 15
Hours
  Day 14: number analyzed (Participants) | 13
  Day 14 | 39.8 (47)
  Day 22 | 42.6 (24)
  Day 31: number analyzed (Participants) | 10
  Day 31 | 33.5 (80)

8. Primary Outcome: Apparent Oral Clearance (CL/F) of Tenofovir Alafenamide (TAF)
Description: Apparent oral clearance of TAF was calculated as "dose/plasma area under the curve (AUC)" on day 14, 22, and 31.
Time Frame: Days 14, 22, and 31
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 20
L/hr
  Day 14: number analyzed (Participants) | 19
  Day 14 | 84.6 (64)
  Day 22 | 52.9 (59)
  Day 31: number analyzed (Participants) | 16
  Day 31 | 100.8 (88)

9. Primary Outcome: Minimum Total Plasma Concentration (Cmin) for Tenofovir Alafenamide (TAF)
Description: Minimum total plasma concentration (Cmin) following a 25mg dose of TAF on day 14, 22, and 31. Cmin for TAF was obtained directly by visual inspection of the plasma concentration versus time profiles over 24 hours postdose.
Time Frame: Days 14, 22, and 31
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 23
ng/mL
  Day 14 | 2.4 (4.5)
  Day 22: number analyzed (Participants) | 22
  Day 22 | 2.9 (6)
  Day 31: number analyzed (Participants) | 16
  Day 31 | 2 (3.1)

10. Primary Outcome: Minimum Total Plasma Concentration (Cmin) for Tenofovir (TFV)
Description: Minimum total plasma concentration (Cmin) following a 25mg dose of tenofovir alafenamide (TAF) on day 14, 22, and 31. Cmin for TFV was obtained directly by visual inspection of the plasma concentration versus time profiles over 24 hours postdose.
Time Frame: Days 14, 22, and 31
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 22
ng/mL
  Day 14 | 9.1 (4.2)
  Day 22: number analyzed (Participants) | 20
  Day 22 | 7.2 (3.2)
  Day 31: number analyzed (Participants) | 15
  Day 31 | 8.7 (4.5)

11. Secondary Outcome: Plasma Area Under the Curve (AUC) for Intracellular Tenofovir Di-phosphate During the Dosing Interval of 0 to 24 Hours (AUC0-24hr)
Description: Plasma area under the curve (AUC) during the dosing interval of 0 to 24 hours (AUC0-24hr) on day 14, 22, and 31 of intracellular tenofovir di-phosphate using the linear-up/log-down trapezoidal rule using noncompartmental methods on Phoenix WinNonlin ®
Time Frame: 0-24 hours post dosing on days 14, 22, and 31
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 23
hr*ng/ml
  Day 14 | NA (NA) — Insufficient drug concentrations above intracellular assay lower limit of quantification (LLOQ)
  Day 22 | NA (NA) — Insufficient drug concentrations above intracellular assay lower limit of quantification (LLOQ)
  Day 31 | NA (NA) — Insufficient drug concentrations above intracellular assay lower limit of quantification (LLOQ)

12. Secondary Outcome: Terminal Half-life (t½) of Intracellular Tenofovir-diphosphate
Description: Half-life calculated as natural log of 2[ ln(2)]/lambda Z of TFV on day 14, 22, and 31.
Time Frame: Days 14, 22, and 31
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 23
Hours
  Day 14 | NA (NA) — Insufficient drug concentrations above intracellular assay lower limit of quantification (LLOQ)
  Day 22 | NA (NA) — Insufficient drug concentrations above intracellular assay lower limit of quantification (LLOQ)
  Day 31 | NA (NA) — Insufficient drug concentrations above intracellular assay lower limit of quantification (LLOQ)

ADVERSE EVENTS:
Time Frame: Up to day 49
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 22/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pharmacokinetic Study in Healthy Volunteers (N=28)
Palpitations (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 2
COVID-19 (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Amylase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 1
Blood bicarbonate decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 5
Blood cholesterol increased (Investigations) | 5
Blood creatine phosphokinase increased (Investigations) | 2
Blood glucose decreased (Investigations) | 1
Blood glucose increased (Investigations) | 3
Blood phosphorus decreased (Investigations) | 4
Blood potassium decreased (Investigations) | 2
Blood sodium decreased (Investigations) | 3
Blood sodium increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 2
C-reactive protein increased (Investigations) | 3
Lipase increased (Investigations) | 6
Low density lipoprotein increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 12
Loss of consciousness (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT03510468/Prot_SAP_000.pdf